CLINICAL TRIAL: NCT02357849
Title: The Role of Antidepressants or Antipsychotics in Preventing Psychosis: Fluoxetine vs Aripiprazole Comparative Trial (FACT)
Brief Title: Fluoxetine vs Aripiprazole Comparative Trial (FACT)
Acronym: FACT
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Christoph U. Correll, MD, Professor of Psychiatry and Molecular Medicine Hofstra North Shore LIJ School of Medicine, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 11-199
Record Dates: First submitted 2014-09-30; First posted 2015-02-06 (Estimated); Results first posted 2023-11-15 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Attenuated Psychosis Syndrome
MeSH Terms: interventions — Aripiprazole; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Active Comparator): To increase homogeneity and assure treatment with a clinically effective dose, patients will undergo a fixed titration phase during the first four weeks (2mg wk1, 5mg wk2, 10mg wk3, 5-30 mg wk4-24), with the option to slow or halt the titration or decrease the target dose if intolerability develops. After 3 weeks, dosing will be flexible and left up to clinical choice and need (5-30mg).
  Interventions: Drug: Aripiprazole
- Fluoxetine (Active Comparator): To increase homogeneity and assure treatment with a clinically effective dose, patients will undergo a fixed titration phase during the first four weeks (5mg wk1, 10mg wk2, 20mg wk3, 10-60mg wk3-24), with the option to slow or halt the titration or decrease the target dose if intolerability develops. After 3 weeks, dosing will be flexible and left up to clinical choice and need(10-60mg).
  Interventions: Drug: Fluoxetine

INTERVENTIONS:
Drug: Aripiprazole — see arm description
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Fluoxetine — see arm description
  Other Names: Prozac
  Arms: Fluoxetine

SUMMARY:
We are conducting a randomized, 24-week, double-blind study, comparing fluoxetine with aripiprazole in 48 patients with attenuated positive symptoms at a level of at least moderate severity.

DETAILED DESCRIPTION:
To Compare Fluoxetine and Aripiprazole on All-cause Discontinuation/Need to Add Another Psychiatric Medication, Symptomatic Improvement, and Adverse Effects

ELIGIBILITY:
Inclusion Criteria:

* consent obtained from patients and their parents (assent for patients under 18);
* age 12-25 years (inclusive);
* English-speaking;
* at least one positive (Scale A) SOPS score of 3-5, i.e., moderate, moderately severe or severe.

Exclusion Criteria:

* lifetime diagnosis of an Axis I psychotic disorder, including: schizophreniform disorder, schizophrenia, schizoaffective disorder, bipolar disorder, or major depression with psychotic features;
* current psychosis (any positive symptom SOPS score of 6, i.e., extreme);
* current diagnosis of Major Depressive Disorder, single episode or recurrent, severe without psychotic features;
* current stimulant treatment;
* history of neurological, neuroendocrine or other medical condition known to affect the brain;
* any significant medical condition that contra-indicates treatment with either aripiprazole or fluoxetine;
* past or current substance dependence; sunstance abuse within the last 4 weeks;
* IQ < 70.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2014-07; Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph U Correll, MD, Principal Investigator — North Shore LIJ
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: outpatient clinic
Groups:
- Aripiprazole: Intervention arm
- Fluoxetine: Active control arm
Period: Overall Study
Arm/Group | Aripiprazole | Fluoxetine
Started | 4 | 5
Completed | 2 | 2
Not Completed | 2 | 3
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Fluoxetine | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.5 (1.3) | 16.0 (1.7) | 15.8 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 1 | 2 | 3
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9
Treatment Failure [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Failure
Description: Time to either all-cause-discontinuation or need to add another psychotropic agent
Time Frame: 24 weeks
Population: Data was not collected
Arm/Group | Aripiprazole | Fluoxetine
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Prodromal Symptoms (SOPS) Total Scores
Description: Change in Prodromal Symptoms (SOPS) total scores (range: 0-30, higher = worse)
Time Frame: 24 weeks
Population: Data was not collected
Arm/Group | Aripiprazole | Fluoxetine
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Patients With Specific Adverse Effects
Description: Number of patients with any adverse effects based on spontaneous report
Time Frame: 24 weeks
Population: Data was not collected
Arm/Group | Aripiprazole | Fluoxetine
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Social and Role Functioning Scores
Description: Change in social and role functioning scores (range: 0-10, higher sores = better outcome)
Time Frame: 24 weeks
Population: Data was not collected
Arm/Group | Aripiprazole | Fluoxetine
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Subjective Well-being Questionnaire
Description: Subjective well-being questionnaire (Total score rang: 20-120, with higher scores indicating greater well-being)
Time Frame: 24 weeks
Population: Data was not collected
Arm/Group | Aripiprazole | Fluoxetine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Aripiprazole | Fluoxetine
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/49/NCT02357849/Prot_SAP_000.pdf
  • Informed Consent Form (2016-09-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT02357849/ICF_001.pdf